CLINICAL TRIAL: NCT07051746
Title: Effectiveness of Metacognitive Training on Symptoms and Cognitive Biases in Taiwanese Individuals With Mental Disorders: A One-Group Pretest-Posttest Study
Brief Title: Effectiveness of Traditional Chinese Metacognitive Training (MCT) in Patients With Schizophrenia, Depression, or Bipolar Disorder Attending a Psychiatric Day Hospital in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZI-YU LIN (Other)
Responsible Party: Sponsor-Investigator, ZI-YU LIN, Principal Investigator, National Taiwan University
Organization: National Taiwan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202506037RIN
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metacognitive Training Group (Experimental): Participants in this arm will receive group-based Metacognitive Training (MCT), the Traditional Chinese version adapted for the Taiwanese population. The intervention consists of 8 sessions delivered twice weekly over 4 weeks. Each session focuses on cognitive biases commonly associated with psychotic and affective disorders, including jumping to conclusions, attribution biases, and social cognitive deficits, etc.
  Interventions: Behavioral: Metacognitive Training (MCT), Traditional Chinese version

INTERVENTIONS:
Behavioral: Metacognitive Training (MCT), Traditional Chinese version — The intervention is a culturally adapted version of Metacognitive Training (MCT) for psychiatric populations in Taiwan. The program consists of 8 group sessions over 4 weeks. Each session includes psychoeducation, cognitive exercises, and group discussion to help participants recognize and reduce cognitive biases.

SUMMARY:
Schizophrenia is characterized by positive symptoms such as delusions and hallucinations, which significantly impact daily functioning. While antipsychotics are the primary treatment, many patients exhibit resistance or intolerance. Metacognitive Training (MCT) has shown promise in addressing cognitive biases related to positive symptoms, offering potential benefits as an adjunct to pharmacological treatment. Additionally, cognitive biases are prevalent in other psychiatric disorders, such as bipolar disorder and major depression, and are closely related to the onset and persistence of emotional symptoms. Preliminary studies have supported the effectiveness of MCT in reducing depressive symptoms and related biases. However, its effects in Taiwan remain unexplored. Therefore, this study aims to examine the effectiveness of the Traditional Chinese version of MCT for individuals with schizophrenia in Taiwan.

This study adopts a one-group pretest-posttest design, recruiting 26 participants to undergo an 8-session MCT group intervention over four weeks. Assessments include the Chinese versions of the Psychotic Symptom Rating Scales (C-PSYRATS), the Traditional Chinese version of the PROMIS Depression and Anxiety Short Forms (4a v1.0), the Modified Davos Assessment of Cognitive Biases Scale (MCL-DACOBS), the Self-reported Graphic Personal and Social Performance Scale (SRG-PSP), Self-Reported Activities of Daily Living Scale, third version (sf-ADLS), and Neuro-QoL Item Bank v2.0 - Cognitive Function- Short Form. Participant satisfaction is also collected. Statistical analyses will utilize non-parametric Wilcoxon Signed-Rank Test and Cohen's d for effect size calculations.

Despite limitations such as a single-group design and recruitment from one hospital, this study is the first to examine MCT's applicability in Taiwanese clinical settings. Expected outcomes include improvements in positive symptoms, depressive and anxiety symptoms, cognitive biases, cognitive functioning, daily living skills, and social functioning. Future research should validate these findings through randomized controlled trials across multiple sites.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Diagnosed with schizophrenia, major depressive disorder, or bipolar disorder based on DSM-5 criteria by a psychiatrist.
* Currently enrolled in a psychiatric day hospital.
* Judged by an occupational therapist as capable of understanding written/spoken Mandarin and completing Chinese-language questionnaires.
* No changes in psychiatric medication within the past month.

Exclusion Criteria:

* History of severe hearing or visual impairments.
* Severe psychiatric symptoms or attention deficits that would prevent full participation in a 60-minute session, as judged by the therapist.
* Presence of inappropriate social behaviors such as aggression, sexual harassment, or antisocial behavior.
* Ongoing major life crises or recent traumatic events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-10-03 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Change in PROMIS Depression 4a T-score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  PROMIS Depression 4a v1.0 (Traditional Chinese version) is a 4-item patient-reported outcome scale. Items are rated 1-5 and converted into T-scores; higher T-scores indicate greater depression severity.
Change in C-PSYRATS Total Score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  The Chinese version of the Psychotic Symptom Rating Scales (C-PSYRATS) includes 17 items measuring severity of delusions and auditory hallucinations. Each item is rated 0-4, with higher scores indicating more severe symptoms.
Change in PROMIS Anxiety 4a T-score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  PROMIS Anxiety 4a v1.0 (Traditional Chinese version) is a 4-item patient-reported scale. Items are rated 1-5 and converted into T-scores; higher T-scores reflect higher anxiety severity.
Change in MCL-DACOBS Total Score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  The Modified Chinese version of the Davos Assessment of Cognitive Biases Scale (MCL-DACOBS) includes 42 items across cognitive biases, limitations, and avoidance. Each item is rated on a 7-point scale; higher scores indicate greater cognitive distortions.

SECONDARY OUTCOMES:
Change in Neuro-QoL Cognitive Function Short Form Score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  The Neuro-QoL Cognitive Function Short Form (Traditional Chinese version) contains 8 self-report items. Each is rated on a 1-5 scale, with higher scores indicating better perceived cognitive function.
Change in SRG-PSP Total Score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  The Self-Reported Graphic version of the Personal and Social Performance Scale (SRG-PSP) assesses role performance, interpersonal relationships, self-care, and disruptive behaviors. Each domain is rated 1-3; higher scores in most domains reflect better function.
Change in sf-ADLS Total Score | Baseline and Week 5 (within 1 week after completing the final MCT session)
  The Self-Reported Activities of Daily Living Scale, 3rd edition (sf-ADLS), includes 14 items rated 1-3. Higher total scores indicate greater independence in daily life.
Participant Satisfaction with Metacognitive Training (MCT) Program | Week 5 (within 1 week after completing the final MCT session)
  A 4-item self-reported questionnaire developed by the investigator to assess participants' satisfaction with the MCT program. Each item is rated on a 4-point scale: 1 = Very Dissatisfied, 2 = Dissatisfied, 3 = Satisfied, 4 = Very Satisfied. The questionnaire evaluates perceived helpfulness, understanding, utility, and overall satisfaction. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Department of Psychiatry, General Psychiatry Day Hospital, Taipei, Taiwan Province, Taiwan